CLINICAL TRIAL: NCT05485090
Title: Cross-cultural Adaptation Into French of the Safety Assessment Scale for Elderly People With a Major Neurocognitive Disorder Living at Home.
Brief Title: Cross-cultural Adaptation of the Safety Assessment Scale for Elderly People With a Major Neurocognitive Disorder Living at Home.
Acronym: ESTRAD
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Other Study IDs: GHRMSA 1209; 2021-A02428-33 (Other: ANSM)
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Major Neurocognitive Disorder
Keywords: Safety; Dementia; Reliability; Validity; Screening
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Phase : Test-Retest Reliability: Caregivers will complete the questionnaire twice with the same investigator. The interval between the two questionnaires is 3 to 10 days.
  Interventions: Other: Questionnaire : Adapted Safety Assessment Scale
- Test Phase : Inter-rater Reliability: Caregivers will complete the questionnaire twice with two different investigators. The interval between the two questionnaires is 3 to 10 days.
  Interventions: Other: Questionnaire : Adapted Safety Assessment Scale

INTERVENTIONS:
Other: Questionnaire : Adapted Safety Assessment Scale — Patients caregivers will complete the questionnaire twice : once at enrollment, then 3 to 10 days after enrollment.

SUMMARY:
The main objective of this study is to adapt the Canadian French version of the safety assessment scale for use in France. The Safety Assessment Scale was developped for community healthcare providers working with elderly people with dementia who are being cared for at home, to assess the risk of accidents. The short version of the Safety Assessment Scale is a screening tool and the longer version provides an in-depth evaluation of safety.

This scale is a risk assessment grid for accidents and injuries at home for elderly people with major neurocognitive disorders, available in English and French (Canadian). There are two versions:

* The short version is used for screening. A score of 11 to 14 indicates a moderate risk of injury, while a score ≥ 15 indicates a high risk of injury;
* The long version is used for in-depth assessment when the score on the short version indicates a moderate or high risk of injury. The questionnaire is divided into nine sections:

  1. Caregiver and environment, 2/smoking, 3/fire and burns, 4/nutrition, 5/food poisoning and toxic substances, 6/medication and health problems, 7/wandering and adaptation to temperature changes, 8/trauma, and 9/driving.

The short version includes some of the questions from sections 1 to 7 of the long version.

DETAILED DESCRIPTION:
Secondary objectives:

The other objectives of this study are to assess the test-retest reliability and the inter-rater reliability of the translated scale and to evaluate the internal consistency of the long version of the translated scale.

Conduct of research:

Caregivers of patients with major neurocognitive disorders included in the study will complete the adapted scale with an investigator. A pre-test phase will be carried out with 10 caregivers: the caregivers will complete the questionnaire only once with an investigator.

After this phase, the translated Safety Assessment Scale will be corrected if there are difficulties in understanding certain words or sentences. The new scale will then be evaluated on two cohorts of 53 caregivers (cohort 1: caregivers will complete the adapted scale twice with the same investigator; cohorte 2: caregivers will complete the adapted scale twice with two different investigators).

ELIGIBILITY:
Inclusion Criteria:

* Patient living at home or hospitalized with a planned return home
* Patient with a major neurocognitive disorder (Diagnostic and Statistical Manual of Mental Disorders, fifth version) :

  * evidence of significant cognitive decline from a previous level of performance in one or more cognitive domains (complex attention, social cognition) based on : a concern by the individual, a knowledgeable informant, or the clinician about a significant decline in cognitive function ; and a deficit in cognitive performance, preferably documented by standardized neuropsychological tests or by another quantified clinical assessment
  * the cognitive deficits interfere with independence in daily activities. At least, assistance should be required with complex instrumental activities of daily living, such as paying bills or managing medications.
  * the cognitive deficits do not occur exclusively in the context of a delirium.
  * the cognitive deficits are not better explained by another mental disorder (e.g., major depressive disorder, schizophrenia).
* Patient with at least one caregiver:

  * reliable (no suspicion of cognitive or psychiatric disorders and/or inappropriate behavior such as manipulation or abuse)
  * able to answer the questionnaire (i.e., knows the patient's lifestyle)
* No objection to participating in the study from the caregiver and the patient (if able to understand the study)
* No objection to guardian participation for patients under guardianship or curatorship

Exclusion Criteria:

* Patient totally socially isolated or without a reliable caregiver
* Bedridden patients
* For hospitalized patients, no planned return home
* Patients under judicial protection

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caregivers of elderly people with a major neurocognitive disorder living at home. Caregivers will be selected by healthcare professionals working in geriatric care.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Test-retest Reliability | 10 days
  The caregiver will complete the questionnaire (adapted Safety Assessment Scale) twice with the same investigator

SECONDARY OUTCOMES:
Inter-rater Reliability | 10 days
  The caregiver will complete the questionnaire (adapted Safety Assessment Scale) twice with two different investigators.
Internal consistency of the long version of the adapted Safety Assessment Scale | 10 days
  The internal consistency of the items will be evaluated within each of the 9 sections of the scale by calculating the Cronbach's alpha coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Clémence BONNOT, Occupational Therapist, Principal Investigator — Groupe Hospitalier de la Region de Mulhouse et Sud Alsace
Locations (1):
- GHRMSA, Mulhouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to the article — https://santepsy.ascodocpsy.org/index.php?lvl=notice_display&id=417792